CLINICAL TRIAL: NCT07343882
Title: Quantification of Systemic Congestion by Ultrasound As a Predictor of Weaning Failure From Mechanical Ventilation
Acronym: SCOUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-CCS-2024-185
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Weaning Failure; Pulmonary Edema - Acute; Mechanical Ventilation; POCUS; VExUS
Keywords: Weaning induced pulmonary edema; Venous Excess Ultrasound grading system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound study (Experimental): Prior to SBT: A complete set of pulmonary, cardiac, and VExUS ultrasounds will be performed and stored for later analysis by blinded experts.
  At the end of SBT: repeat pulmonary and cardiac ultrasounds
  Interventions: Diagnostic Test: point of care ultrasound

INTERVENTIONS:
Diagnostic Test: point of care ultrasound — Complete set of pulmonary, cardiac, and VExUS ultrasounds

SUMMARY:
Mechanical ventilation is an essential, life-saving therapy in the ICU, allowing critically ill patients to rest and recover. Transitioning patients back to spontaneous breathing-known as weaning-is clinically challenging. The first attempt, the Spontaneous Breathing Trial (SBT), fails in 10-30% of cases. Identifying the mechanisms behind failure is crucial, as unsuccessful weaning prolongs ICU stay and increases the risk of reintubation, which worsens prognosis. The SCOUT study aims to improve prediction and management of weaning failure.

The main objective of the study is to evaluate whether a specific ultrasound-based method, the Venous Excess Ultrasound Score (VExUS), can predict failure of weaning from mechanical ventilation. A key pathophysiological factor is systemic venous congestion. When a patient initiates an SBT, the increased respiratory effort shifts venous return and may precipitate cardiovascular decompensation with pulmonary fluid accumulation, termed weaning-induced pulmonary edema (WIPO). Notably, this may occur even in patients without known cardiac disease.

Detecting clinically relevant congestion before SBT is difficult. Fluid balance and body weight are imprecise, physical examination lacks sensitivity, and biomarkers such as NT-proBNP have limited predictive capacity. VExUS offers a promising, non-invasive approach by directly assessing venous flow patterns in major veins (inferior vena cava, hepatic, portal, and renal veins), providing an estimation of systemic venous pressure and congestion. The central hypothesis is that elevated VExUS grades prior to SBT will identify patients at high risk of failure, enabling proactive optimization and potentially improving outcomes.

SCOUT is designed as a prospective, multicenter, observational study. Standard clinical management of mechanical ventilation and weaning remains unchanged. After informed consent, baseline data will be obtained immediately before SBT, including vital signs, ventilator parameters, blood sampling, and three non-invasive ultrasound assessments: cardiac, pulmonary, and VExUS. During the 30-120-minute SBT, the patient breathes with reduced ventilatory support while their clinical tolerance is evaluated. At the end of the SBT, selected measurements are repeated. Weaning failure is defined as: early termination of SBT due to intolerance, need for invasive or non-invasive ventilation within 48 h after extubation, or death within 48 h. Data are anonymized and stored securely (REDCap) in compliance with Spanish and EU data protection regulations.

The study is low-risk and provides no direct individual benefit, but may benefit future ICU patients by improving weaning strategies and prognostication.

DETAILED DESCRIPTION:
1. Protocol overview and Rationale Weaning patients from invasive mechanical ventilation represents a significant daily challenge within the intensive care unit (ICU). The process is complex, and failure can lead to prolonged ventilation, increased morbidity, and worsened patient outcomes. The "Quantification of Systemic Congestion by Ultrasound As a Predictor of Weaning Failure from Mechanical Ventilation (SCOUT)" study is a prospective investigation designed to evaluate a novel, non-invasive method for identifying patients at high risk of weaning failure before a trial is even attempted.

   The core clinical problem addressed by this study is the high incidence of weaning failure, which occurs in 10-30% of patients. While respiratory complications are a common cause, up to 30% of failures are attributed to cardiovascular origins. A key mechanism in these cases is systemic congestion, which can lead to weaning-induced pulmonary edema (WIPO). This condition occurs when the physiological stress of a spontaneous breathing trial (SBT) causes a rapid shift of fluid into the central circulation, overwhelming cardiac capacity and flooding the lungs, even in patients without a prior history of heart failure.

   Current methods for assessing a patient's fluid status and risk of congestion have significant limitations. Clinicians often rely on metrics such as cumulative fluid balances, daily weight changes, physical examination findings, and biomarkers. However, these tools have proven to be insufficiently reliable or specific for accurately predicting which patients will develop WIPO during an SBT. While tools like echocardiography are useful for diagnosing pulmonary edema after it has already occurred, they have not demonstrated utility in identifying at-risk patients beforehand. Similarly, pulmonary ultrasound can detect lung edema (B-lines) but not identify high risk patients before it occurs.

   This study will investigate the Venous Excess Ultrasound (VExUS) grading system as a predictive tool. VExUS is a novel, point-of-care ultrasound protocol that provides a comprehensive assessment of systemic venous congestion. It integrates ultrasound measurements of the inferior vena cava with Doppler flow patterns in the hepatic veins, portal vein, and intrarenal veins to generate a score that quantifies the degree of venous congestion.

   Given that systemic congestion is a central mechanism in WIPO, a tool that can reliably measure it at the bedside holds immense potential. VExUS provides real-time, repeatable information, allowing for dynamic patient monitoring. The central justification for this study is that by using the VExUS score to assess a patient before initiating an SBT, clinicians may be able to identify those at high risk of cardiovascular-related weaning failure. This proactive identification would allow for targeted therapeutic measures to be implemented preemptively, thereby improving a patient's readiness for weaning, reducing the likelihood of failure, and minimizing the consequences associated with prolonged mechanical ventilation. This clinical rationale underpins the study's formal hypotheses and objectives.
2. Study Hypotheses and Objectives

   * Primary Hypothesis: The assessment of systemic congestion using the VExUS ultrasound score immediately prior to a SBT can identify patients who are at risk of weaning failure.
   * Primary Objective: To evaluate the utility of the VExUS score for predicting the failure of weaning from mechanical ventilation.

   Secondary Hypotheses and Objectives

   - Secondary Hypotheses: The VExUS score demonstrates superior diagnostic performance in identifying patients at risk of SBT failure compared to other methods (pulmonary ultrasound, cardiac ultrasound, and biomarkers).

   Patients with a higher VExUS score before the SBT experience a longer total weaning duration.

   The assessment of systemic congestion via VExUS can predict the need for reintubation.

   - Secondary Objectives: To compare the diagnostic performance of different methods (biomarkers, pulmonary ultrasound, cardiac ultrasound) for predicting SBT failure.

   To evaluate whether a correlation exists between the VExUS-assessed degree of congestion and the number of days required for weaning.
3. Study Design and Methodology The study is designed as a prospective, multicenter registry. The design is considered quasi-experimental because it evaluates the effect of an intervention, the comprehensive ultrasound assessment, on a cohort of patients.

   - Study Population and Sample Size

   Inclusion Criteria:

   Patients aged > 18 years. Admitted to an Intensive Care Unit (ICU). Requiring invasive mechanical ventilation for more than 48 hours. Meeting the center's standard criteria to begin weaning and undergo an SBT.

   Exclusion Criteria:

   Inadequate ultrasound window for assessment. Presence of "do not reintubate" orders. Patients with a tracheostomy. Presence of atrial fibrillation. Diagnosed liver cirrhosis (portal hypertension). Absence of qualified personnel to perform the ultrasound at the time of the SBT.

   Denial of informed consent.

   - Sample Size: The study requires a total of 350 patients for the final analysis. This calculation is based on an assumed 30% weaning failure rate, an alpha risk of 0.05, and a statistical power greater than 0.8. The enrollment target will be higher to account for an estimated 20% loss to follow-up.

   The following sequence of procedures and data collection will be applied to each enrolled patient.

   At Study Inclusion The following baseline variables will be collected:
   * Demographic data (age, sex, patient history).
   * Reason for ICU admission and for initiation of mechanical ventilation.
   * Severity scores (SAPS III and APACHE II).
   * Duration of mechanical ventilation prior to the first SBT.

   Prior to SBT initiation A comprehensive set of measurements will be performed immediately before the trial begins:
   * Vital Signs and Ventilator Parameters: Heart rate, blood pressure, respiratory rate, support level, tidal volume, FiO2, and PEEP.
   * Analytical Parameters: Arterial blood gases (pH, O2, CO2), and the most recent laboratory results for renal function, liver function, electrolytes, and ProBNP.
   * Ultrasound Assessments: A complete set of pulmonary, cardiac, and VExUS ultrasounds will be performed and stored for later analysis by blinded experts.

   The SBT will be conducted according to each center's protocol, lasting between 30 and 120 minutes via T-tube or pressure support. Immediately before the patient is reconnected to the ventilator (in case of failure) or extubated (in case of success), a second set of measurements will be taken, including vital signs, an arterial blood gas sample, Pro-BNP level, and repeat pulmonary and cardiac ultrasounds.

   Definition of Weaning Failure Weaning failure, the primary study outcome, is defined as either a failure of the spontaneous breathing trial or a failure of extubation.Failure of the Spontaneous Breathing Trial: The SBT is interrupted due to clinical intolerance, requiring reconnection to the ventilator. Extubation Failure: The patient requires rescue with invasive or non-invasive mechanical ventilation within 48 hours of extubation, or the patient dies within 48 hours of extubation.

   At ICU Discharge The final variables to be collected include:
   * Fluid balance from admission to the day of the SBT.
   * Total fluid balance
   * Total duration of mechanical ventilation, including the number of days from the first SBT to final extubation, and ICU/hospital length of stay.
   * Patient status (alive/dead) at ICU discharge, 30 days post-discharge, and 90 days post-discharge.
4. Data Management and Quality Assurance The study will utilize a custom database designed in the RedCap application at the coordinating center, Hospital de la Santa Creu i Sant Pau. This system is fully compliant with all applicable data protection regulations. Upon completion of the study, the database will be irreversibly anonymized to protect participant confidentiality.

   The General Coordinating team holds responsibility for monitoring data quality across all participating centers. This process includes a random review of 5% of participants from each center to control for data accuracy and completeness.

   The Coordinating Team will issue automated alerts to investigators to recover any missing information. To ensure the integrity of the final dataset, any participant with missing primary variables or more than 10% of missing secondary variables will be excluded from the final analysis.

   Each site's principal investigator is responsible for ensuring that the data entered into the electronic Case Report Form (CRF) is accurate and consistent with source documents, such as patient medical records. Investigators must agree to provide direct access to these source documents for monitoring, auditing, and inspection by ethics committees or regulatory authorities upon request.
5. Statistical Analysis Plan

   - Data Presentation Qualitative Variables: Data will be summarized as absolute numbers and corresponding percentages.

   Quantitative Variables: Data will be presented as mean and 95% interval confidence, or as median and interquartile range for non-normally distributed variables. The Kolmogorov-Smirnov test will be used to assess data distribution.

   - Comparative Analysis Group Comparisons: Differences between groups will be analyzed using the Student's t-test, χ2 test, or Mann-Whitney U test, as appropriate for the data type and distribution.

   Paired Comparisons (pre- vs. post-SBT): Measurements taken before and after the SBT will be compared using a paired Student's t-test or a Wilcoxon signed-rank test, depending on data distribution.

   Predictive Performance Analysis To address the primary objective, Receiver Operating Characteristic (ROC) curve analysis will be employed to evaluate the ability of VExUS and other methods to predict weaning failure. The optimal threshold value for each predictive index will be determined using the Youden index, which maximizes the sum of sensitivity and specificity. The non-parametric DeLong method will be used to formally compare the areas under the ROC curves for different predictors.

   Software All statistical analyses will be conducted using the SPSS v25 and Stata software packages.
6. Acknowledged Protocol Limitations

   * Operator-Dependence of Ultrasound: Ultrasound assessments are inherently operator-dependent, meaning that results can vary based on the skill and technique of the person performing the scan. The protocol mitigates this by requiring all assessments to be performed by trained personnel, but inter-observer variability remains a potential limitation.
   * Heterogeneity of Pre-SBT Care: While the protocol standardizes the SBT procedure itself, the clinical management of patients on mechanical ventilation leading up to the SBT may differ between participating centers. This variability in pre-trial care introduces a potential confounding factor that could influence patient outcomes.
   * Inherent VExUS Limitations: The VExUS score itself has known limitations, as certain clinical conditions can influence its measurements and alter the results. Although the protocol addresses most of these through its detailed exclusion criteria, they represent a limitation of the tool itself that must be considered when interpreting the findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years.
* Admitted to an Intensive Care Unit (ICU).
* Requiring invasive mechanical ventilation for more than 48 hours.
* Meeting the center's standard criteria to begin weaning and undergo an SBT.

Exclusion Criteria:

* Inadequate ultrasound window for assessment.
* Presence of "do not reintubate" orders.
* Patients with a tracheostomy.
* Presence of atrial fibrillation.
* Diagnosed liver cirrhosis (portal hypertension).
* Absence of qualified personnel to perform the ultrasound at the time of the SBT.
* Denial of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Weaning failure | From the start of the spontaneous breathing trail to 48 hours after
  The primary objective of the SCOUT study is: To evaluate the utility of VExUS to predict weaning failure from mechanical ventilation.
  Defining the Weaning Failure
  A patient is considered to have met the primary outcome if they experience any one of the following events:
  * The Spontaneous Breathing Trial (SBT) is interrupted due to clinical intolerance, requiring reconnexion to mechanical ventilation.
  * The patient is extubated but requires rescue with mechanical ventilation (either invasive or non-invasive) within the subsequent 48 hours.
  * The patient is extubated and dies within the subsequent 48 hours.
Utility of the VExUS score for predicting the failure of weaning from mechanical ventilation | From the start of the spontaneous breathing trial to the next 48 hours
  The primary objective of the SCOUT study is: To evaluate the utility of VExUS to predict weaning failure from mechanical ventilation.
  The Venous Excess Ultrasound Score (VExUS) is expressed as four grades (0-3):
  VExUS 0: No congestion VExUS 1: Mild congestion VExUS 2: Moderate congestion VExUS 3: Severe congestion
  A patient is considered to have met the primary outcome (weaning failure) if they experience any one of the following events:
  * The Spontaneous Breathing Trial (SBT) is interrupted due to clinical intolerance, requiring reconnexion to mechanical ventilation.
  * The patient is extubated but requires rescue with mechanical ventilation (either invasive or non-invasive) within the subsequent 48 hours.
  * The patient is extubated and dies within the subsequent 48 hours.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Background] Ferre A, Guillot M, Lichtenstein D, Meziere G, Richard C, Teboul JL, Monnet X. Lung ultrasound allows the diagnosis of weaning-induced pulmonary oedema. Intensive Care Med. 2019 May;45(5):601-608. doi: 10.1007/s00134-019-05573-6. Epub 2019 Mar 12. PMID 30863935
- [Background] Zapata L, Vera P, Roglan A, Gich I, Ordonez-Llanos J, Betbese AJ. B-type natriuretic peptides for prediction and diagnosis of weaning failure from cardiac origin. Intensive Care Med. 2011 Mar;37(3):477-85. doi: 10.1007/s00134-010-2101-4. Epub 2010 Dec 9. PMID 21152896
- [Background] Zapata L, Suarez-Montero JC, Lopez-Garzon PA. Association between diastolic dysfunction and fluid balance in critically ill patients during weaning from mechanical ventilation. Med Intensiva (Engl Ed). 2023 Dec;47(12):708-716. doi: 10.1016/j.medine.2023.05.012. Epub 2023 Jun 26. PMID 37380508
- [Background] Vignon P. Cardiopulmonary interactions during ventilator weaning. Front Physiol. 2023 Sep 7;14:1275100. doi: 10.3389/fphys.2023.1275100. eCollection 2023. PMID 37745230
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740